CLINICAL TRIAL: NCT00000253
Title: Effects of Nitrous Oxide: A Dose-Response Analysis
Brief Title: Effects of Nitrous Oxide: A Dose-Response Analysis - 5
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Double
Other Study IDs: NIDA-08391-5; R01DA008391 (NIH); R01-08391-5
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Opioid-Related Disorders; Substance-Related Disorders
Keywords: nitrous oxide; inhalant; subjective effects; healthy volunteer
MeSH Terms: conditions — Opioid-Related Disorders; Substance-Related Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- Placebo + 10% N2O (Active Comparator): 0% N2O inhaled during psychomotor testing, 10% N2O inhaled during psycho motor testing, then subject's choice of the 2.
  Interventions: Drug: 10% N2O
- Placebo + 20% N2O (Active Comparator): Placebo inhaled during psychomotor testing, 20% N2O inhaled during psychomotor testing, then subject's choice of the 2.
  Interventions: Drug: 20% N2O
- Placebo + 30% N2O (Active Comparator): Placebo inhaled during psychomotor testing, 30% N2O inhaled during psychomotor testing, then subject's choice of the 2.
  Interventions: Drug: 30% N2O
- Placebo + 40% N2O (Active Comparator): Placebo inhaled during psychomotor testing, 40% N2O inhaled during psychomotor testing, then subject's choice of the 2.
  Interventions: Drug: 40% N2O

INTERVENTIONS:
Drug: 10% N2O
  Arms: Placebo + 10% N2O
Drug: 20% N2O
  Arms: Placebo + 20% N2O
Drug: 30% N2O
  Arms: Placebo + 30% N2O
Drug: 40% N2O
  Arms: Placebo + 40% N2O

SUMMARY:
The purpose of this study is to conduct experiments to examine subjective and reinforcing effects of nitrous oxide. Mood altering and psychomotor effects will be tested on non-drug abusers and preference procedures will be used to assess reinforcing effects. To examine the subjective, psychomotor, and reinforcing effects of nitrous oxide in healthy volunteers. This is a dose-response analysis.

ELIGIBILITY:
Please contact site for information.

Ages: 21 Years to 37 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 1994-11; Primary Completion 1996-03 (Actual); Study Completion 1996-03 (Actual)

PRIMARY OUTCOMES:
Choice of N2O vs. placebo | After each pair of sample tests
  Subjects underwent 4 sessions consisting of 2 sample tests (inhaling placebo and inhaling varying doses of N2O), then choosing which inhalant they wanted for a choice test. The subject & the technician administering the inhalant were blinded. During each intervention and each session, subjects underwent psychomotor testing.

CONTACTS AND LOCATIONS:
Overall Officials: James Zacny, Ph.D., Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Anesthesia & Critical Care, Chicago, Illinois, United States

REFERENCES:
- [Background] Behavioral Pharmacology, 1996, 7: 194-199.